CLINICAL TRIAL: NCT00971295
Title: Effect of Eslicarbazepine Acetate on the Pharmacokinetics of Metformin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-125
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Neuropathic Pain
Keywords: eslicarbazepine acetate; zebinix; metformin
MeSH Terms: conditions — Neuralgia | interventions — Metformin; eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence A (Experimental): Eslicarbazepine acetate + Metformin period followed by washout period followed by Metformin period
  Interventions: Drug: Metformin; Drug: Eslicarbazepine acetate
- Treatment Sequence B (Experimental): Metformin period followed by washout period followed by Eslicarbazepine acetate + Metformin period
  Interventions: Drug: Metformin; Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Metformin — 850 mg metformin hydrochloride, once as oral single-dose and once after pre-treatment with once-daily dose of ESL 1200 mg for 6 days
  Other Names: Glucophage
Drug: Eslicarbazepine acetate
  Other Names: Zebinix

SUMMARY:
The primary objective was to investigate whether multiple-dose administration of eslicarbazepine acetate affects the pharmacokinetics of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or who smoke ≤ 10 cigarettes or equivalent per day.
* Able and willing to give written informed consent.
* (If female) Not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) Negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* History of relevant atopy or drug hypersensitivity.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to each treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Used medicines within 2 weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion.
* Used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Participated in more than 2 clinical trials within the 12 months prior to screening.
* Donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or with medical dietary restrictions.
* Could not communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to give written informed consent.
* (If female) Pregnant or breast-feeding.
* (If female) Of childbearing potential and she did not use an approved effective contraceptive method (double-barrier or intra-uterine device) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, MD, PhD, Principal Investigator — BIAL - Portela & Ca, S.A
Locations (1):
- Human Pharmacology Unit (UFH)Section of Clinical Research (SIC), Department of Research & Development (DID), BIAL - Portela & Cª, SA,, Mamede Do Coronado, Portugal

REFERENCES:
- [Result] Rocha JF, Vaz-da-Silva M, Almeida L, Falcao A, Nunes T, Santos AT, Martins F, Fontes-Ribeiro C, Macedo T, Soares-da-Silva P. Effect of eslicarbazepine acetate on the pharmacokinetics of metformin in healthy subjects. Int J Clin Pharmacol Ther. 2009 Apr;47(4):255-61. doi: 10.5414/cpp47255. PMID 19356391

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: Treatment Sequence A:
  Eslicarbazepine acetate + Metformin period followed by washout period followed by Metformin period
  850 mg metformin hydrochloride, 1200 mg ESL
- Treatment Sequence B: Treatment Sequence B:
  Metformin period followed by washout period followed by Metformin + Eslicarbazepine acetate
  850 mg metformin hydrochloride, 1200 mg ESL
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Metformin + ESL: Metformin HCl 850 mg, ESL 1200 mg
  Metformin + eslicarbazepine: 850 mg metformin hydrochloride, once as oral single-dose and once after pre-treatment with once-daily dose of ESL 1200 mg for 6 days
Arm/Group | Metformin + ESL
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Maximum Observed Plasma Metformin Concentration
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Metformin: Metformin HCl 850 mg
Arm/Group | Metformin + ESL | Metformin
Number analyzed (Participants) | 20 | 19
ng/mL | 1091 (27.6) | 1224 (21.9)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Description: time of occurrence of maximum observed plasma metformin concentration
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Metformin + ESL | Metformin
Number analyzed (Participants) | 20 | 19
hours | 2.66 (46.9) | 2.53 (40.4)

3. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration From Time Zero to Infinity
Description: area under the plasma metformin concentration from time zero to infinity
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Metformin + ESL | Metformin
Number analyzed (Participants) | 20 | 19
ng*h/mL | 7362 (26.7) | 7688 (21.4)

ADVERSE EVENTS:
Arm/Group | Metformin + ESL | Metformin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + ESL (N=20) | Metformin (N=20)
Erythropapular rash (Skin and subcutaneous tissue disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Constipation (General disorders) | 1 | 0
Herpes labialis (Infections and infestations) | 0 | 1
Right forearm ecchymosis (General disorders) | 1 | 0
Recurrent vasovagal reaction (Nervous system disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilateral popliteal erythromacular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Eczema aggravated (Skin and subcutaneous tissue disorders) | 1 | 0
Acute gastroenteritis (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Eyelid hematoma (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes